CLINICAL TRIAL: NCT00034216
Title: Biospecimen Acquisition From Human Subjects
Brief Title: Collection of Blood From Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020179; 02-C-0179
Record Dates: First submitted 2002-04-24; First posted 2002-04-24 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-11-06

CONDITIONS: Prostate Cancer; Breast Cancer; Colon Cancer; Lung Cancer; Liver Cancer
Keywords: Suppressor Cells; T-cells; CD4+ / CD25+ cells; Natural History; Cancer; Malignancy; Blood Sample
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy volunteers 18 years of age and older
- Participants: Participants with cancer 18 years of age and older

SUMMARY:
This study will collect blood from patients with cancer to study the level of cells which decrease the immune response (suppressor cells) before and after chemotherapy. Patients 18 years of age and older with cancer may participate. This study does not involve treatment.

Participants will have about 50 ml (3 tablespoonfuls) of blood drawn. Depending on their condition, patients may be invited to enroll in a clinical research study involving chemotherapy, radiotherapy, or surgery. Additional 40-ml blood samples may be drawn during the course of treatment.

DETAILED DESCRIPTION:
Background:

* Correlative studies performed on biospecimens of human subjects can be used to investigate the biology of solid tumors, inform the development of new strategies for treating those cancers, and evaluate these new therapeutic approaches. Specific areas of interest include, but are not limited to:
* the underlying mechanisms of tumor-specific immune response and suppression in cancer patients
* genetic and molecular profiling of tumors through circulating tumor cell (cTC), circulating DNA, and tissue analysis
* investigation of potential early diagnostic and prognostic indicators for solid tumors such as cTCs and miRNA expression of serum exosomes
* identification of mechanisms of drug-related adverse events and correlation with clinical parameters
* the role of commensal gut microbiota in both the innate and adaptive responses to tumors as well as with the use of anticancer agents

Objectives:

* Analyze biospecimens such as tissue, urine, saliva, stool and blood components, which include serum, leukocytes, peripheral blood mononuclear cells (PBMC), and circulating tumor cells (cTC), of human subjects.
* Correlate analysis results with clinical parameters such as demographics, toxicities, and treatment outcomes.
* Undertake genetic analysis of both prokaryotic and eukaryotic samples for advanced mutational analysis.

Eligibility:

* Patients and healthy volunteers whose biospecimens are of interest to NIH investigators.
* 18 years of age or older.

Design:

- Cases will be evaluated by NCI or Interventional Radiology, NIH Clinical Center personnel. Blood, tissue, urine, saliva or other samples may be collected at the initial visit and at follow-up visits.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with a known or suspected malignancy and healthy volunteers 18 years of age and older are eligible.

Performance status of ECOG 0, 1, 2, or 3 for admission to this protocol.

Ability to understand and the willingness to sign a written informed consent document.

INCLUSION FOR APHERESIS:

Note: Effective with Amendment CC, participants will no longer be asked to undergo apheresis. This content is being retained for historical reference.

Hemoglobin greater than or equal to 10 mg/dL and platelet count > 75,000/mm(3)

Weight greater than 25 kg

HIV negative

Prothrombin Time - within normal limits

Partial Thromboplastin Time - within normal limits

Medically indicated central line in place or adequate peripheral venous access

EXCLUSION CRITERIA:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary clinical; healthy volunteers may include NIH employees
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Estimated)
Dates: Start 2002-07-16 (Actual)

PRIMARY OUTCOMES:
Undertake genetic analysis of both prokaryotic and eukaryotic samples for advanced mutational analysis. | ongoing
  Undertake genetic analysis of both prokaryotic and eukaryotic samples for advanced mutational analysis.
Correlate analysis results with clinical parameters such as demographics, toxicities, and treatment outcomes. | ongoing
  Correlate analysis results with clinical parameters such as demographics, toxicities, and treatment outcomes.
Collection of tissue, urine, saliva, stool and blood components, which include serum, leukocytes, peripheral blood mononuclear cells (PBMC), and circulating tumor cells (cTC), of human subjects. | ongoing
  Analyze tissue, urine, saliva, stool and blood components, which include serum, leukocytes, peripheral blood mononuclear cells (PBMC), and circulating tumor cells (cTC), of human subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Marte, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-C-0179.html